CLINICAL TRIAL: NCT03274518
Title: Expanded Hemodialysis Versus Online Hemodiafiltration: a Pilot Study on Intradialytic Hemodynamics and Fluid Status
Brief Title: Expanded Hemodialysis Versus Online Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Caldin da Silva, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16928
Record Dates: First submitted 2017-08-08; First posted 2017-09-07 (Actual); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Dialysis Related Complication; Dialysis Hypotension; Hemodialysis-Induced Symptom
Keywords: Hemodialysis; Hemodiafiltration; fluid status; hemodynamics

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator who collects laboratorial, hemodynamics and bioimpedance data will be blinded for intervention (online hemodiafiltration or expanded hemodialysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Hemodiafiltration (Active Comparator): The olHDF technique combines diffusion with high convection rates in which the dialysis fluid, free of toxins and pyrogens, is used to prepare the replacement fluid.
  The online module of dialysis machine prepares the replacement fluid by a cold sterilization process. There is a cross-flow water preparation, in order to avoid the accumulation of possible contaminants. The addition of bicarbonate and acid solutions to water follows the process. Next, the ready-for-infusion dialysis solution is passed through another ultrafilter prior to being infused into patients.
  Interventions: Device: Online Hemodiafiltration
- Expanded Hemodialysis (Experimental): More recently, membranes with high cutoff values, but with tight pore size distribution have been developed. The main concept is to keep both cutoff and retention onset values close to each other, but with a cutoff value lower than of albumin. This should allow removal of middle-to-high weight range uremic toxins, with very low albumin leak. Thus, these membranes, denominated high retention onset (HRO) membranes, allow performing both diffusive and convective processes in a conventional hemodialysis machine.
  Interventions: Device: Expanded Hemodialysis

INTERVENTIONS:
Device: Expanded Hemodialysis — Intervention: Conversion from conventional HD to expanded hemodialysis por 1 month.
  High cutoff with high retention onset dialyzers allow clearance of middle molecules, without reducing significantly serum concentration of albumin. It allows higher convective clearance in comparison to conventional hemodialysis, but it is unknown if such clearance is similar to online hemodiafiltration. Therefore, the aim of the present intervention is to compare this dialyzer with online hemodiafiltration
  Other Names: Theranova Dialyzer
  Arms: Expanded Hemodialysis
Device: Online Hemodiafiltration — Intervention: Conversion from conventional HD to online Hemodiafiltration por 1 month.
  Online hemodiafiltration has been associated with lower incidence of intradialytic hypotension in comparison to conventional hemodialysis.
  Arms: Online Hemodiafiltration

SUMMARY:
Conventional hemodialysis (HD) is essential for the treatment of end-stage renal disease (ESRD) patients, by reducing serum concentration of uremic toxins and correcting fluid overload.

Nevertheless, HD removes almost exclusively low-range uremic toxins. Therefore, medium-range molecules, such as beta-2-microglobulin might accumulate in tissues, leading to many clinical complications, such as neuropathies, tendinopathies, anemia, bone mineral disease and reduced growth in children.

Convective methods might reduce incidence of these complications, by removing molecules of medium-range molecular weight. Online hemodiafiltration (olHDF) is the most extensively used method in this regard. Nevertheless, there are some barriers to the wider introduction of this method in clinical practice, since specific machines are needed for this procedure, the costs with dialysis lines are higher and water consumption increases. More recently, the development of new membranes for hemodialysis allowed removal of medium- and high-range uremic toxins, with albumin retention. Thus, they allow removal of a broad range of uremic toxins, without changing dialysis machine or increasing water consumption. Such therapy is known as expanded hemodialysis (HDx).

The aim of this present study is to compare the extraction of middle-size molecules, the hemodynamic behavior, fluid and nutritional status of patients submitted to olHDF or HDx, in a crossover study.

DETAILED DESCRIPTION:
Hypothesis

Our hypothesis is that HDx is noninferior to olHDF in the following parameters:

* Hemodynamic stability
* Nutritional and fluid status
* Removal of beta-2 microglobulin

Objectives To evaluate each patient, through a prospective, randomized and cross-over study, the intradialytic hemodynamic behavior, fluid and nutritional status assessed by electrical bioimpedance and B2M removal in two dialytic modalities: HDFol versus HDx.

Concise methods

1. Clinical and laboratorial data Clinical data will be collected from the institution's chart, recorded and filled with all necessary precautions to keep confidentiality of patient's information. They are: baseline renal disease, age, history of smoking, sedentary lifestyle, presence of comorbidities such as hypertension and diabetes mellitus, family history of cardiovascular disease, history of coronary and cerebrovascular disease and medications.

   Laboratory tests used to determine the biochemical, hematological and bone mineral profile characteristics will be obtained from routinely collected exams. Such exams are processed by the Central Laboratory of Hospital das Clínicas / FMUSP.
2. Dialysis All dialysis procedures will be performed by the Dialog+ Admea™ machine (BBraun Melsungen AG, Germany).

   The olHDF will be prescribed as follows: blood flow 350 - 400 ml/min, dialysate flow 800 ml/min, post-dilution flow (90-100 ml/min), with high-flux Xevonta™ (BBraun Melsungen AG, Germany) or CAHP/DICE™ (Baxter Healthcare Corporation, Germany) dialyzers, with surface area of 1.7-2.4 m². The duration of each session will be from 3,5h to 4h, depending on current dialysis prescription. Total substitution volume will be higher than 20 L per session.

   HDx will follow the same prescription of olHDF, regarding blood and dialysate flows and dialysis duration. There will be no substitution volume. Theranova™ dialyzers (Baxter Healthcare Corporation, Germany) will be used for each session.

   Before initiating protocol and during the washout period, patients will be submitted to high-flux HD, which is the standard treatment in our service.
3. Hemodynamic monitoring Cardiac output index (CI), stroke volume (SV - integrated mean of the flow waveform between the current upstroke and the dichotic notch), peripheral arterial resistance (PAR - ratio of mean arterial pressure to stroke volume multiplied by heart rate) and blood pressure (BP) will be accessed by finger beat to-beat monitor Finometer™ (Finapress Medical Systems BV, Arnhem, The Netherlands), within 15 minutes after starting olHDF or HDx sessions (predialysis) and again, 15 minutes before its end (post-dialysis).
4. Bioelectrical impedance Segmental tetrapolar bioelectrical impedance (BIS) will be performed in all patients while recumbent, before starting study protocol and before each phase of the study (HDx or olHDF), by the multifrequency InBody™ S10 (Biospace Co., Ltd., Korea) device. It allows assessment of the following parameters regarding body fluids: total body water, total extracellular body water, lower limbs total water content, lower limbs extracellular water content. Additionally, α-angle, which is a marker of cellular integrity and nutritional status, will be noted.
5. Blood and Effluent samples Blood samples will be collected pre-session, mid-session and post-dialysis sessions, both in the first and last dialysis sessions of each of the periods studied (HDFol or HDx). Pre-session blood samples will be collected immediately after arteriovenous fistula puncture and the middle and post-session samples will be collected from the arterial line, 2 minutes after reduction of blood flow to 50 ml/min and suspension of dialysate flow and/ or replacement.

In addition, partial and homogeneous collection of the effluent will be performed by a drainage hose, with an infusion pump operating continuously at a rate of 1l/h. The whole effluent of dialysis session will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are on maintenance hemodialysis at Hospital das Clínicas and agree to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Patients who cannot understand or who refuse to sign the informed consent form; Patients who are currently on daily hemodialysis or online hemodiafiltration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno C Silva, PhD, Principal Investigator — Renal Division, Unversity of São Paulo
Locations (1):
- Hospital das Clínicas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karohl C, de Paiva Paschoal J, de Castro MC, Elias RM, Abensur H, Romao JE Jr, Passlick-Deetjen J, Jorgetti V, Moyses RM. Effects of bone remodelling on calcium mass transfer during haemodialysis. Nephrol Dial Transplant. 2010 Apr;25(4):1244-51. doi: 10.1093/ndt/gfp597. Epub 2010 Jan 29. PMID 20118484
- [Result] Cheng YL, Shek CC, Wong FK, Choi KS, Chau KF, Ing TS, Li CS. Determination of the solute removal index for urea by using a partial spent dialysate collection method. Am J Kidney Dis. 1998 Jun;31(6):986-90. doi: 10.1053/ajkd.1998.v31.pm9631843.
- [Result] Alvares VRC, Ramos CD, Pereira BJ, Pinto AL, Moyses RMA, Gualano B, Elias RM. Pneumatic Compression, But Not Exercise, Can Avoid Intradialytic Hypotension: A Randomized Trial. Am J Nephrol. 2017;45(5):409-416. doi: 10.1159/000471513. Epub 2017 Apr 14. PMID 28407637
- [Result] Cheng YL, Shek CC, Wong AK, Wong FK, Chau KF, Li CS. A partial dialysate collection method. Int J Artif Organs. 1997 Jan;20(1):14-7. PMID 9062826
- [Result] Argiles A, Ficheux A, Thomas M, Bosc JY, Kerr PG, Lorho R, Flavier JL, Stec F, Adele C, Leblanc M, Garred LJ, Canaud B, Mion H, Mion CM. Precise quantification of dialysis using continuous sampling of spent dialysate and total dialysate volume measurement. Kidney Int. 1997 Aug;52(2):530-7. doi: 10.1038/ki.1997.364. PMID 9264013
- [Result] Oliveira CM, Kubrusly M, Mota RS, Silva CA, Choukroun G, Oliveira VN. The phase angle and mass body cell as markers of nutritional status in hemodialysis patients. J Ren Nutr. 2010 Sep;20(5):314-20. doi: 10.1053/j.jrn.2010.01.008. Epub 2010 Mar 19. PMID 20303790
- [Result] Silva BC, Freitas GR, Silva VB, Abensur H, Luders C, Pereira BJ, de Oliveira RB, Castro MC, Moyses RM, Elias RM. Hemodynamic behavior during hemodialysis: effects of dialysate concentrations of bicarbonate and potassium. Kidney Blood Press Res. 2014;39(5):490-6. doi: 10.1159/000368459. Epub 2014 Nov 23. PMID 25532082
- [Result] Silva BC, Moyses RM, Silva VB, Freitas GR, Elias RM. Parathyroidectomized patients have impaired capacity of peripheral vascular constriction during hemodialysis. Hemodial Int. 2016 Jan;20(1):50-5. doi: 10.1111/hdi.12309. Epub 2015 Apr 28. PMID 25923250
- [Result] Jimenez ZN, Silva BC, Reis LD, Castro MC, Ramos CD, Costa-Hong V, Bortolotto LA, Consolim-Colombo F, Dominguez WV, Oliveira IB, Moyses RM, Elias RM. High Dialysate Calcium Concentration May Cause More Sympathetic Stimulus During Hemodialysis. Kidney Blood Press Res. 2016;41(6):978-985. doi: 10.1159/000452601. Epub 2016 Dec 16. PMID 27978518

RESULTS

PARTICIPANT FLOW:
Groups:
- Online Hemodiafiltration: Arm description: Online Hemodiafiltration first, then expanded hemodialysis.
  First, patients changed fom conventional HD to online hemodiafiltration for 1 month.
  Then, patients returned to conventional HD for 2 weeks (washout period). Then, patients underwent the second intervention (expanded hemodialysis) for 1 month, in a cross-over design.
- Expanded Hemodialysis: Arm description: expanded hemodialysis first, then online hemodiafiltration.
  Intervention: Conversion from conventional HD to expanded hemodialysis for 1 month.
  Then, patients returned to conventional HD for 2 weeks (washout period). Then, they underwent the second intervention (online hemodiafiltration), for 1 month, in a cross-over design.
Period: First Intervention
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Started (First intervention: online hemodiafiltration, for 30 days) | 8 | 8 (First intervention: expanded hemodialysis, for 30 days.)
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Started (Patients returned from online Hemodiafiltration to conventional hemodialysis for 15 days.) | 8 | 8 (Patients returned from expanded hemodialysis to conventional hemodialysis for 15 days.)
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Started (Second intervention: patients from this group underwent expanded hemodialysis for 30 days.) | 8 | 8 (Second intervention: patients from this group underwent online hemodiafiltration for 30 days.)
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Online Hemodiafiltration: Patients were included in this study group per sequence:
  Online hemodiafiltration (olHDF) first for 1 month, then expanded hemodialysis (HDx) for 1 month.
  Baseline characteristics assessed:
  * Age
  * Gender
  * Ethnicity
  * Region of Enrollment
  * Serum Beta-2 Microglobulin
- Expanded Hemodialysis: Patients were included in this study group per sequence:
  Expanded hemodialysis (HDx) first for 1 month, then online hemodiafiltration (olHDF) for 1 month.
  Baseline characteristics assessed:
  * Age
  * Gender
  * Ethnicity
  * Region of Enrollment
  * Serum Beta-2 Microglobulin
- Total: Total of all reporting groups
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39.5 [28.7 to 43.5] | 46 [28.7 to 59.5] | 39.5 [28.7 to 52.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 8 | 8 | 16
Serum Beta-2 Microglobulin [Mean (Standard Deviation); unit: mcg/ml] | 23.2 (6.9) | 27.8 (5.5) | 25.2 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Medium Molecule Clearance
Description: Beta-2-Microglobulin clearance
Time Frame: One month after starting protocol
Population: Beta-2 Microglobulin clearance (ml/min)
Measure: Median (Inter-Quartile Range); unit: ml/min
Groups:
- Expanded Hemodialysis: High cutoff with high retention onset dialyzers allow clearance of middle molecules, without reducing significantly serum concentration of albumin.
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Number analyzed (Participants) | 16 | 16
ml/min | 53 [41.8 to 63.7] | 59.5 [50.5 to 70]
Statistical Analysis 1: Comparison: Online Hemodiafiltration vs Expanded Hemodialysis; Test type: Non-Inferiority — The non-inferiority margin was defined as difference within 20% in comparison to reference method (olHDF); p = 0.4534, t-test, 2 sided

2. Primary Outcome: Medium Molecule Removal
Description: Beta-2-Microglobulin extraction
Time Frame: One month after starting protocol
Population: Beta-2-microglobulin mass extraction (mg)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Number analyzed (Participants) | 16 | 16
mg | 198 (81) | 239 (86)
Statistical Analysis 1: Comparison: Online Hemodiafiltration vs Expanded Hemodialysis; Test type: Non-Inferiority — The non-inferiority margin was defined as difference within 20% in comparison to reference method (olHDF); p = 0.1179, t-test, 2 sided

3. Secondary Outcome: Intradialytic Hemodynamics
Description: noninvasive cardiac output assessment
Time Frame: Cardiac output (liters per minute) one month after starting protocol
Population: Intradialytic cardiac output variation (post-pre dialysis), l/min
Measure: Median (Inter-Quartile Range); unit: l/min
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Number analyzed (Participants) | 16 | 16
l/min | -1.3 [-2.2 to -0.3] | -1.4 [-3 to -1.1]
Statistical Analysis 1: Comparison: Online Hemodiafiltration vs Expanded Hemodialysis; Test type: Non-Inferiority — The non-inferiority margin was defined as difference within 20% in comparison to reference method (olHDF); p = 0.3054, t-test, 2 sided

4. Other Pre Specified Outcome: Fluid Status
Description: noninvasive assessment of extracellular and total body water
Time Frame: One month after starting protocol
Measure: Mean (Standard Deviation); unit: liter/liter
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
Number analyzed (Participants) | 16 | 16
liter/liter | 0.39 (0.01) | 0.385 (0.01)
Statistical Analysis 1: Comparison: Online Hemodiafiltration vs Expanded Hemodialysis; Test type: Non-Inferiority — The lower the ECW/TBW ratio, the lower pre-dialysis excess fluid. A non-inferiority margin was defined as difference within 10% from reference method (olHDF); p = 0.045, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Description: No adverse events noted
Groups:
- Online Hemodiafiltration: The olHDF technique combines diffusion with high convection rates in which the dialysis fluid, free of toxins and pyrogens, is used to prepare the replacement fluid.
  The online module of dialysis machine prepares the replacement fluid by a cold sterilization process. There is a cross-flow water preparation, in order to avoid the accumulation of possible contaminants. The addition of bicarbonate and acid solutions to water follows the process. Next, the ready-for-infusion dialysis solution is passed through another ultrafilter prior to being infused into patients.
  Online Hemodiafiltration: Intervention: Conversion from conventional HD to online Hemodiafiltration por 1 month.
  Online hemodiafiltration has been associated with lower incidence of intradialytic hypotension in comparison to conventional hemodialysis.
- Expanded Hemodialysis: More recently, membranes with high cutoff values, but with tight pore size distribution have been developed. The main concept is to keep both cutoff and retention onset values close to each other, but with a cutoff value lower than of albumin. This should allow removal of middle-to-high weight range uremic toxins, with very low albumin leak. Thus, these membranes, denominated high retention onset (HRO) membranes, allow performing both diffusive and convective processes in a conventional hemodialysis machine. Expanded Hemodialysis: Intervention: Conversion from conventional HD to expanded hemodialysis por 1 month.
  High cutoff with high retention onset dialyzers allow clearance of middle molecules, without reducing serum concentration of albumin. It allows higher convective clearance in comparison to conventional hemodialysis, but it is unknown if such clearance is similar to online hemodiafiltration. Therefore, the aim of the present intervention is to compare this dialy
Arm/Group | Online Hemodiafiltration | Expanded Hemodialysis
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The sample size was small and trial length was relatively short. We did not directly assessed albumin extraction. Besides, the relatively low ultrafiltration coefficient of both dialyzers limited dialysis performance in all treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03274518/Prot_SAP_002.pdf
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03274518/ICF_003.pdf